CLINICAL TRIAL: NCT02137057
Title: The Effect of Spinal Anesthesia on Heart Rate Variability in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0167
Record Dates: First submitted 2014-05-11; First posted 2014-05-13 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Heart Rate Variability; Diabetes; Spinal Anesthesia
Keywords: Heart Rate Variability; spinal anesthesia; DM; cardiac autonomic dysfunction
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control ( patients without diabetes): patients without diabetes
- DM ( patients with diabetes): patients with diabetes

SUMMARY:
Cardiac autonomic neuropathy is a common complication of diabetes and is associated with resting tachycardia. Regional anesthesia could interrupt normal autonomic activity by central sympathetic blockade. The investigators evaluate the relation of severity of diabetes and heart rate variability, also the impact of spinal anesthesia on the change of heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing lower limb surgery with spinal anesthesia (ASA class 1,2,3)

Exclusion Criteria:

* severe coagulopathy, short height, arrhythmia patients, patients taken medication which could affect autonomic nervus system (bata- blocker or alpha-blocker)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing lower limb surgery with spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change of Heart rate variability during spinal anesthesia : total power, power of LF and HF, and LF/HF ratio | 10 min before spinal anesthesia (T0: Baseline ) 10 min (T1), 20 min (T2) and 30 min (T3) after spinal injection

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Lee SH, Lee DH, Ha DH, Oh YJ. Dynamics of heart rate variability in patients with type 2 diabetes mellitus during spinal anaesthesia: prospective observational study. BMC Anesthesiol. 2015 Oct 8;15:141. doi: 10.1186/s12871-015-0125-6. PMID 26450424